CLINICAL TRIAL: NCT02834169
Title: French National Registry of Rare Peritoneal Surface Malignancies (RENAPE Registry)
Brief Title: French National Registry of Rare Peritoneal Surface Malignancies
Acronym: RENAPE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0406
Record Dates: First submitted 2016-06-30; First posted 2016-07-15 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Rare Peritoneal Surface Malignancies; Pseudomyxoma Peritonei; Peritoneal Mesothelioma; Desmoplastic Small Round Cell Tumor; Psammocarcinoma; Primary Peritoneal Serous Carcinoma; Diffuse Peritoneal Leiomyomatosis; Appendiceal Mucinous Neoplasms
Keywords: Rare peritoneal surface malignancies; pseudomyxoma peritonei; peritoneal mesothelioma; desmoplastic small round cell tumor; psammocarcinoma; primary peritoneal serous carcinoma; diffuse peritoneal leiomyomatosis; appendiceal mucinous neoplasms; registry; population-based database
MeSH Terms: conditions — Pseudomyxoma Peritonei; Desmoplastic Small Round Cell Tumor; Cystadenocarcinoma, Serous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- pseudomyxoma peritonei: Data from pseudomyxoma peritonei cases will be used to generate descriptive statistics on demographics, clinical characteristics including prevalence and incidence of co-morbidities, treatment patterns, and patient outcomes (resulting from treatment or disease).
  Interventions: Other: Non interventional
- peritoneal mesothelioma: Data from peritoneal mesothelioma cases will be used to generate descriptive statistics on demographics, clinical characteristics including prevalence and incidence of co-morbidities, treatment patterns, and patient outcomes (resulting from treatment or disease).
  Interventions: Other: Non interventional
- desmoplastic small round cell tumor: Data from desmoplastic small round cell tumor cases will be used to generate descriptive statistics on demographics, clinical characteristics including prevalence and incidence of co-morbidities, treatment patterns, and patient outcomes (resulting from treatment or disease).
  Interventions: Other: Non interventional
- psammocarcinoma: Data from primary peritoneal serous carcinoma cases will be used to generate descriptive statistics on demographics, clinical characteristics including prevalence and incidence of co-morbidities, treatment patterns, and patient outcomes (resulting from treatment or disease).
  Interventions: Other: Non interventional
- primary peritoneal serous carcinoma: Data from primary peritoneal serous carcinoma cases will be used to generate descriptive statistics on demographics, clinical characteristics including prevalence and incidence of co-morbidities, treatment patterns, and patient outcomes (resulting from treatment or disease).
  Interventions: Other: Non interventional
- diffuse peritoneal leiomyomatosis: Data from diffuse peritoneal leiomyomatosis cases will be used to generate descriptive statistics on demographics, clinical characteristics including prevalence and incidence of co-morbidities, treatment patterns, and patient outcomes (resulting from treatment or disease).
  Interventions: Other: Non interventional
- appendiceal mucinous neoplasms: Data from appendiceal mucinous neoplasms cases will be used to generate descriptive statistics on demographics, clinical characteristics including prevalence and incidence of co-morbidities, treatment patterns, and patient outcomes (resulting from treatment or disease).
  Interventions: Other: Non interventional

INTERVENTIONS:
Other: Non interventional — Data collection

SUMMARY:
Despite advances in the management of and changes in clinical practice, little is known about the epidemiology, patterns of care and outcomes of rare peritoneal surface malignancies patients in France.

In order to better understand the characteristics of rare peritoneal surface malignancies and to evaluate treatment strategies, the RENAPE registry aims at the collection of data from patients presenting with a rare peritoneal surface malignancy in France. Data will be entered prospectively in a specifically designed and secured web database.

All RENAPE's centres and physicians are invited to register patients with a rare peritoneal surface malignancy diagnosis and to participate to the registry. Data will be evaluated within regular time frames, focusing on types of rare peritoneal surface malignancies, treatment modalities and patient outcomes (e.g. survival, recurrence), thereby contributing to the better understanding of these rare cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible if they have a histologically proven rare peritoneal surface malignancy.

Exclusion Criteria:

* Histological diagnostic of peritoneal surface malignancy not confirmed
* Expected clinical follow up data not available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospectively or retrospectively diagnosed patients with rare peritoneal surface malignancies.
Sampling Method: Non-Probability Sample
Enrollment: 2171 (Actual)
Dates: Start 2010-10; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of rare peritoneal surface malignancies | year 5
  Collect detailed clinical and histological diagnosis for estimating annual incidence rate

SECONDARY OUTCOMES:
Impact of specific treatment strategies | year 5
  Collect detailed therapeutic strategies (surgical procedure, chemotherapy, etc.) on patients with rare peritoneal surface malignancies

CONTACTS AND LOCATIONS:
Overall Officials: François-Noël GILLY, Prof, Principal Investigator — Hospices Civils de Lyon - Centre Hospitalier Lyon Sud - Service de Chirurgie Générale et Digestive - 165 chemin du grand Revoyet, PIERRE-BENITE, FRANCE, 69495
Locations (33):
- France (33):
  - Institut de Cancérologie de l'Ouest - Paul Papin, Angers
  - CHU Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - CHU Estaing, Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand
  - AP-HP Louis MOURIER, Colombes
  - CHU Bocage, Dijon
  - CHU A. Michallon, La Tronche
  - Centre Oscar Lambret, Lille
  - CHRU Claude Huriez, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital La Timône, Marseille
  - Institut du Cancer Montpellier, Montpellier
  - CHU Nantes Hôtel-Dieu, Nantes
  - CHU L'Archet II, Nice
  - Institut Curie, Paris
  - AP-HP St Antoine, Paris
  - AP-HP La Pitié-Salpêtrière, Paris
  - AP-HP Lariboisière, Paris
  - AP-HP Hôpîtal Europeen Georges Pompidou, Paris
  - Hospices Civils de Lyon - Centre Hospitalier Lyon Sud - Service de Chirurgie Générale et Digestive - 165 chemin du grand Revoyet,, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - Hôpital Robert Debré, Reims
  - CHU Charles Nicolle, Rouen
  - CHU Nord, Saint-Etienne
  - Institut Cancérologie de l'Ouest - René Gauducheau, Saint-Herblain
  - CHRU Hautepierre, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Hôpital Purpan, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Villeneuve L, Passot G, Glehen O, Isaac S, Bibeau F, Rousset P, Gilly FN; RENAPE Network. The RENAPE observational registry: rationale and framework of the rare peritoneal tumors French patient registry. Orphanet J Rare Dis. 2017 Feb 17;12(1):37. doi: 10.1186/s13023-017-0571-y. PMID 28212684
- See also: Related Info — http://www.renape-online.fr/
- See also: Related Info — https://epidemiologie-france.aviesan.fr/fr/epidemiologie-france/fiches/registre-national-des-tumeurs-rares-du-peritoine
- See also: Related Info — http://www.e-cancer.fr/Professionnels-de-sante/L-organisation-de-l-offre-de-soins/Prise-en-charge-des-cancers-rares/Une-organisation-en-centres-experts